CLINICAL TRIAL: NCT04072328
Title: Propofol vs. Midazolam With Propofol for Sedative Endoscopy in Patients With Previous Paradoxical Reaction to Midazolam
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DongGuk University (Other)
Responsible Party: Principal Investigator, Dong Kee Jang, Assistant Professor, DongGuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2018-02-011
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Sedation; Endoscopy
Keywords: Midazolam; Propofol; Sedation
MeSH Terms: interventions — Propofol; Midazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol alone (Experimental): Participants who receive propofol alone during sedative endoscopy.
  Interventions: Drug: Propofol
- Midazolam with propofol (Active Comparator): Participants who receive midazolam + propofol during sedative endoscopy.
  Interventions: Drug: Propofol; Drug: Midazolam

INTERVENTIONS:
Drug: Propofol — Propofol will be given 0.5 mg/kg bolus initially, and can be administered additionally after a least 30 secs if necessary.
Drug: Midazolam — midazolam with propofol
  Arms: Midazolam with propofol

SUMMARY:
This study is to compare propofol vs. midazolam with propofol for sedative endoscopy in patients with previous paradoxical reaction to midazolam. Patients who meet eligibility criteria will randomly assigned to propofol group or midazolam with propofol group. Then they will receive a sedative endoscopy with close monitoring. The primary outcome is the prevalence of paradoxical response during endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* History of midazolam-induced paradoxical response

Exclusion Criteria:

* Failed to obtain informed consent
* Pregnant or breast feeding women
* A severe cardiopulmonary or vascular disease with symptoms
* Cognitive or mental impairment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
The prevalence of paradoxical response | At the end of endoscopy
  The proportion of participants who show paradoxical response during endoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee TH, Lee CK, Park SH, Lee SH, Chung IK, Choi HJ, Cha SW, Moon JH, Cho YD, Hwangbo Y, Kim SJ. Balanced propofol sedation versus propofol monosedation in therapeutic pancreaticobiliary endoscopic procedures. Dig Dis Sci. 2012 Aug;57(8):2113-21. doi: 10.1007/s10620-012-2234-0. Epub 2012 May 22. PMID 22615018
- [Result] Tae CH, Kang KJ, Min BH, Ahn JH, Kim S, Lee JH, Rhee PL, Kim JJ. Paradoxical reaction to midazolam in patients undergoing endoscopy under sedation: Incidence, risk factors and the effect of flumazenil. Dig Liver Dis. 2014 Aug;46(8):710-5. doi: 10.1016/j.dld.2014.04.007. Epub 2014 Jun 2. PMID 24893689
- [Result] Mancuso CE, Tanzi MG, Gabay M. Paradoxical reactions to benzodiazepines: literature review and treatment options. Pharmacotherapy. 2004 Sep;24(9):1177-85. doi: 10.1592/phco.24.13.1177.38089. PMID 15460178